CLINICAL TRIAL: NCT04585945
Title: Pregnancy Outcomes During the Pandemic: Using Placental Pathology and Gene Expression to Understand Fetal Risk
Brief Title: COVID-19 on Placental Gene Expression and Pathology
Acronym: PROSPER
Status: Completed | Type: Observational
Sponsor: Prisma Health-Upstate (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00101090
Record Dates: First submitted 2020-09-17; First posted 2020-10-14 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: COVID-19; SARS-CoV-2 Infection
MeSH Terms: conditions — COVID-19 | interventions — Gene Expression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Placental specimens for transcriptomic analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group 1 (Cases): Patients that test positive for SARS-CoV-2 infection during pregnancy, including at the time of delivery.
  Interventions: Diagnostic Test: Positive for SARS-CoV-2 infection
- Group 2 (Control): Historic group of patients delivering prior to the COVID-19 pandemic.

INTERVENTIONS:
Diagnostic Test: Positive for SARS-CoV-2 infection — Patients that have a positive test for SARS-CoV-2 infection during pregnancy, including at the time of delivery.
  Groups: Group 1 (Cases)

SUMMARY:
Little is known regarding the effect of antenatal COVID-19 on pregnancy outcomes. The purpose of this study is to determine of COVID-19 alters histopathology and gene expression of the placenta, as evidenced by analysis at time of delivery. The analysis will aim to identify whether resulting abnormal placental pathology or altered metabolism is associated with severity of symptoms (specifically pneumonia, or need for admission), gestational age at onset, and/or placenta efficiency. Histological and gene expression analysis of the placental post-delivery will determine if COVID-19 alters overall placental structure, vascularization, and/or the transcriptome.

DETAILED DESCRIPTION:
The current outbreak of COVID-19, the disease caused by severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), shares similarities to the severe acute respiratory syndrome (SARS) disease outbreak (2002 - 2003) and the ongoing Middle East respiratory syndrome (MERS) outbreak which originated in 2012. All three infections present with a cough, fever, and the potential for lower respiratory tract disease. While SARS and MERS maintain a higher case fatality rate (CFR), the higher transmissibility for COVID-19 results in larger number of cases and deaths. Severe respiratory infections which commonly result in pneumonia, such as SARS and influenza A H1N1, are associated with an increased risk for maternal mortality and stillbirth. Although current evidence does not suggest a higher maternal risk of infection than the general population, little is known on the impact of the infection on pregnancy and adverse neonatal outcomes. A systematic review of Coronavirus spectrum infections reported an 11% increase rate of perinatal death. The exact mechanisms of perinatal deaths are not well characterized.

While there is little evidence to date that suggests SARS-CoV-2 infection is vertically transmissible to the fetus, angiotensin-converting enzyme 2 (ACE2), the confirmed receptor for SARS-CoV-2, has been detected at high levels in the early human placenta and presents with tissue specific activity patterns. Villous cytotrophoblast and syncytiotrophoblast cells exhibit high levels of ACE2 expression during the first trimester while expression in the extravillous trophoblast layer starts low during early pregnancy and then peaks around 24 weeks gestation. Disruption in the vascularization and/or metabolic capacity of the placenta could result in placental insufficiency and suboptimal fetoplacental growth and development. A prior study on placental findings from patients with COVID-19 demonstrated an increase in decidual arteriopathy and patterns of maternal vascular malperfusion (MVM), many of whom were asymptomatic from COVID-19. Additionally, a portion of patients with COVID-19 during pregnancy will experience pneumonia and subsequent hypoxia. We hypothesize that exposure to hypoxemia and maternal respiratory failure may further threaten metabolic demands of the fetoplacental unit during gestation.

Our primary research hypothesis is that COVID-19 disease impacts placental development and function and is mediated by severity and duration of illness. We hypothesize that the impact on placental development will subsequently increase adverse fetal outcomes.

This is a case control research project that will utilize patient data (including chart history) and placental specimens collected from Greenville Memorial Hospital between June 2020 and June 2021 during the COVID-19 outbreak. Controls will be matched using banked placental and cord blood specimens collected at Greenville Memorial Hospital or Northshore University Health system prior to emergence of the COVID-19 outbreak, between March 2017 and December 2019. We plan to use banked samples given the potentially high rate of asymptomatic cases. At the conclusion of the study, samples and data collected at Greenville Memorial Hospital will be deidentified and combined with samples collected at NorthShore University Health Center for subsequent analysis and publication.

Potentially eligible patients will be identified during their routine prenatal care at the Prisma Health OB/GYN Center, through the Prisma Health COVID-19 Registry, or when they are admitted to Greenville Memorial Hospital for delivery. Patients will be evaluated for eligibility based on a review of the medical record. Patients identified prior to hospital admission may be consented at their next prenatal care visit at the OB/GYN Center, Maternal-Fetal Medicine Unit, or when they arrive at Greenville Memorial for delivery. Patients identified as eligible prior to hospital admission for delivery will be marked as eligible under the research tab in their chart. Patients identified prior to hospital admission may be consented and enrolled at their next prenatal care visit at the OB/GYN Center, Maternal-Fetal Medicine Unit, or when they arrive at Greenville Memorial for delivery.

At enrollment, patients will answer a short questionnaire regarding demographics and COVID symptoms. At time of delivery, placental samples and umbilical cord blood will be collected for molecular and histologic assessments of inflammation. Trained nursing, resident, and/or research staff will collect and process these specimens. Because villi develop clonally, gene expression may cluster spatially. To minimize the influence of these variations, staff will obtain 0.4 cm3 biopsies from four separate cotyledons in each placenta and suspend the tissue in a stabilizing agent (AllProtect Tissue Reagent, Qiagen). Deidentified placental biopsies will be batched and shipped to Dr. Greg Miller's laboratory at NorthShore University, Chicago, Illinois, where they will be prepped for analysis involving placental transcription regulation. De-identified placental specimens will be shipped to the UCLA Social Genomics Core, who will measure transcriptional regulation as reflected in the expression of mRNA and miRNA. From de-identified samples, Core technicians will extract RNA using Qiagen RNeasy Mini Kits, and perform QA/QC checks with an Agilent TapeStation. 500 ng of RNA will be converted to cDNA (Illumina TruSeq Stranded Total RNA RiboZero Globin) and sequenced on an Illumina HiSeq 4000 instrument, using protocols that optimally detect mRNA and miRNA. > 50 million sequence reads per sample will be mapped to the RefSeq human genome (hisat2/stringtie) and normalized to transcript counts per million mapped reads for each currently annotated mRNA and miRNA. A trained pathologist at Greenville Memorial will conduct a gross examination of the placenta and prepare cassettes for later histologic evaluation. Deidentified placental slides will be obtained from the pathology lab and will be shipped to NorthShore where a perinatal pathologist will confirm pathology findings. Specifically, hematoxylin and eosin-stained, 5 μm thick sections of the membranes, basal plate, and villous parenchyma will be examined for evidence of both acute and chronic inflammatory lesions in the placenta's three major compartments: membranes, villous parenchyma, and basal plate. The perinatal pathologist at Northshore will additionally examine the placental tissue for COVID using immunohistochemical stains for COVID-19. Medical charts will be abstracted for pregnancy outcomes and complications. Specifically, we will abstract obstetric and medical history, including parity, history of health problems and birth outcomes, body mass index prior to pregnancy, results of oral glucose tolerance tests and gestational diabetes screens, diagnoses of diabetes, hypertension, preeclampsia, and infectious diseases during current pregnancy. Delivery data will include method of delivery and duration of labor, as well as fetal sex, weight, length, and gestational age. Two coders, blind to other data, will abstract each record, and resolve discrepancies by consensus. Once the specified data are collected, no further inquiries into medical records will be performed. In other words, we do not plan to continue abstracting information about mother's or children's health as time goes on. Should we desire to begin doing so, we would seek guidance from the IRB about how to obtain proper consent from participants to do so. We anticipate the study to take place over 1 year. Participants will be involved at the time of their delivery, and their medical records will be reviewed from pregnancy to up to 6 weeks following delivery.

ELIGIBILITY:
Inclusion Criteria:

1. COVID-19 infection during pregnancy, including at time of delivery
2. Age >=18 years
3. ≥13 6/7 weeks' GA

Exclusion Criteria:

1. Known major fetal chromosomal abnormality
2. Other major infection during pregnancy (specifically influenza A or B, cytomegalovirus, toxoplasma, rubella, syphilis, HIV)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population for the present study includes all women delivering at Greenville Memorial Hospital. The opportunity for enrollment may be extended to women that deliver at Greenville Memorial even if they conducted prenatal care outside of the Prisma OB/GYN Center if they meet the eligibility. We aim to recruit 40 patients for analysis. Additionally, 60 samples will be recruited from women delivering at NorthShore Health System who test positive for COVID-19 during pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2020-08-04 (Actual); Primary Completion 2021-04-21 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Inflammatory biomarkers in umbilical cord blood between women with COVID-19 disease in the first, second and third trimester of pregnancy and determine if differences are mediated by severity of the illness. | At the time of delivery.
  Umbilical cord blood will be analyzed using an inflammatory biomarker panel (TNF, IL6, CRP, IL4, IL13)
Differences in placental pathology (inflammatory processes, vasculopathy, and villous maturity) for women with COVID-19 disease and determine of differences are mediated by gestational age at infection or severity of illness. | At the time of delivery.
  A perinatal pathologist will review placental pathology findings to determine the occurrence of inflammatory processes, vasculopathy, and villous maturity, as reflected in histology.
Differences in gene expression analysis for women with COVID-19 disease and determine if differences are medicated by gestational age at infection or severity of illness. | At the time of delivery.
  Gene expression analysis will be conducted to identify altered gene expression patterns related to placental development (inflammation, vascularity, and metabolism).

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Britt, PhD, Principal Investigator — Prisma Health-Upstate
Locations (1):
- Prisma Health Upstate, Greenville, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No